CLINICAL TRIAL: NCT03351517
Title: Preemptive Tapentadol on Post-operative Analgesia Following Total Knee Arthroplasty: A Randomized Double Blind Placebo-controlled Trial.
Brief Title: Preemptive Tapentadol on Post-operative Analgesia Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr Debasish Hota, Prof and Head of the Department, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T/IM-NF/Pharma/02/17
Record Dates: First submitted 2017-11-11; First posted 2017-11-24 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tapentadol arm (Experimental): Single dose of 100 mg of extended release oral tapentadol will be administered 1 hour before surgery.
  Interventions: Drug: Tapentadol 100 MG
- Placebo arm (Placebo Comparator): A comparable placebo will be administered 1 hour before surgery.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tapentadol 100 MG — 100 mg of oral extended release tapentadol will be given to the patients undergoing total knee replacement surgery on spinal anesthesia to evaluate its efficacy in the management of post-operative pain.
  Arms: Tapentadol arm
Drug: Placebo Oral Tablet — A matching placebo will be given to the patients undergoing total knee replacement surgery on spinal anesthesia to evaluate its efficacy in the management of post-operative pain.
  Arms: Placebo arm

SUMMARY:
The study intends to evaluate the efficacy of Tapentadol against placebo as a preemptive analgesic in the management of post-operative pain in the patiens undergoing total knee arthroplasty.

The primary objective is to evaluate th epain score in visual analogue scale at various time points within 24 hours post operarively

DETAILED DESCRIPTION:
METHODOLOGY

* Consent: Participants will be explained the benefit and harm of joining the study and the freedom of withdrawing from the study at any moment they would like to. A full voluntary written informed consent will be obtained from each participant. Study will be conducted following the principles of Helsinki after getting written permission of the institutional ethics committee. Before enrolment of first subject in this study registration for clinical trial will be done.
* Participants: Patients of either sex, above 18 yrs. of age undergoing Total Knee Arthroplasty will be the participants in this study.

  1. Inclusion Criteria:
* Patients both males and females undergoing elective total knee replacement surgery
* Patients are capable to provide an informed consent
* Age 18-75 yrs.

  2. Exclusion Criteria:
* Patients with Asthma, COPD or any other respiratory disease.
* Persistent nausea and vomiting at the time of randomization.
* Epilepsy.
* Treated with mono amine oxidase inhibitors, tricyclic antidepressants, serotonin norepinephrine re uptake inhibitors.
* Patients with ASA grading 3 or more.
* Drug abuse history.
* Opioid tolerance or opioid dependence.
* Renal disease(creatinine>1.5 mg/dl).
* Liver disease (total bilirubin>1.5 mg/dl).
* Known history of opioid allergies.
* Major psychiatric disorder.
* Pregnancy and lactation.
* Emergency surgery.
* Bone tumor
* Migraine patients or patients complaining dizziness, vertigo.

Screening: The trial will be comprised of complete medical history and physical examination and screening. Pre-operative laboratory investigations will be recorded in case record form.

* Randomization: A total of 90 Participants will be selected by computer generated random list.
* Blinding: The study will be conducted in a double blinded manner.
* Treatment Administration and baseline follow up: The participants will be assigned to receive 100 mg of Tapentadol or a matched placebo orally 1 hr before spinal anesthesia in a double-blind manner. All the participants, both control and Tapentadol group will be anesthetized (SP) as per the standard protocol after similar pre-medication. Single dose of injection Paracetamol 1 gm i.v. will be provided in both the groups immediately after operation.
* Assessment of efficacy and safety and Duration: All the subjects will be assessed for pain at rest, before surgery, at 0, 6 12 &, 24 hrs. post operatively by visual analogue scale score(VAS) (0 mm: no pain,100 mm: Worst pain imaginable).16 and TOTPAR SCALE(None-Mild-Moderate-Severe) *. They also will be evaluated for nausea, vomiting, drowsiness, and pruritus and will be rated on0,6,12, & 24 hrs.16. Total rescue analgesic consumption also will be assessed at 24 hrs post operatively 16. The time of 1st request for supplemental analgesia also will be recorded. A blood sample will be obtained from each participant at 0 hrs. post operatively to measure the tapentadol concentration and Cholecystokinin by ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex undergoing elective tota knee replacement surgery
* Patients are capable to provide an informed consent
* Age 18-65 years

Exclusion Criteria:

* Patients with Asthma, copd or any other respiratory disease
* Persistent nausea , vomiting at the time of randomization
* Treated with MAO inhibitors, Tricyclic antidepressants, SSRIs and SNRIs
* Patients with ASA grading 3 or more
* Drug abuse history, opioid tolerance or dependence, known history of opiod allergies
* Renal or liver disease
* Major psychiatric disorder
* Pregnancy and lactation
* Emergency surgery
* Bone tumor, epilepsy or patients with migraine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Assessment of Change of Pain score compared to plecebo by visual analogue scale | 24 hrs. post-operatively( 0,2,4,6,12,24 hrs post operatively)
  All the subjects will be assessed for pain at various time points post-operatively by visual analogue scale(VAS) (minimum value 00- no pain to maximum value-100 - worst pain imaginable) Higher values indicate worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: DEBASISH HOTA, MD,DM, Principal Investigator — AIIMS Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India